CLINICAL TRIAL: NCT07130643
Title: Single-arm Exploratory Study of Efficacy and Safety of CDK4/6 Inhibitors Combined With Endocrine Therapy in HR+/HER2- Neoadjuvant Therapy for Early Breast Cancer
Brief Title: Efficacy and Safety of CDK4/6 Inhibitors Combined With Endocrine Therapy in HR+/HER2- Neoadjuvant Therapy for Early Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xinhong Wu, PhD (Other)
Responsible Party: Sponsor-Investigator, Xinhong Wu, PhD, PhD, Hubei Cancer Hospital
Organization: Hubei Cancer Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-209
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-12

CONDITIONS: HR+/HER2- Breast Cancer
Keywords: neoadjuvant; HR+/HER2- breast cancer; CDK4/6 inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): CDK4/6 inhibitors+Endocrine Therapy every 28 days for 6 cycles
  Interventions: Drug: CDK4/6 inhibitors+Endocrine Therapy

INTERVENTIONS:
Drug: CDK4/6 inhibitors+Endocrine Therapy — CDK4/6 inhibitors：dalpiciclib,palbociclib,abemaciclib,ribociclib

SUMMARY:
This is a single arm, open label, phase 2 trial aimed to investigate the effects and safety of neoadjuvant CDK4/6 inhibitors in combination with endocrine for HR+/HER2- breast cancer. A total of 40 patients with stage II-III HR+/HER2- breast cancer will be enrolled. Six 4-week cycles of adjuvant therapy will be administrated.Premenopausal or perimenopausal patients should combine ovarian function suppression, including bilateral oophorectomy or treatment with gonadotropin-releasing hormone agonists.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old.

  2. Premenopausal and postmenopausal women or men with stage II-III disease (multifocal and/or multifocal early invasive breast cancer) if all tumors on histopathological examination meet the pathological criteria for ER and/or PR > 10% and HER2- (HER2 expression of 0 or 1+ or 2+ and negative FISH test).

  3.Patients had to have histologically confirmed ER and (or PR>10%, HER2 -, early-stage invasive disease.

  4.Intolerance or insensitivity to neoadjuvant chemotherapy: 2 cycles of neoadjuvant chemotherapy, PD/SD according to tumor evaluation, old age, and basic diseases can not tolerate chemotherapy.

  5. ECOG PS score 0-2.

  6. Patients must be able and willing to swallow and retain oral medications.

  7. In premenopausal women, a serum or urine pregnancy test had to be negative within 14 days of enrollment or in women who had been amenorrhea for less than 12 months at enrollment.

  8.Patients who had received neoadjuvant endocrine therapy were eligible if they were enrolled within 6 months of the initial histologic diagnosis and had completed no more than 2 months of neoadjuvant endocrine therapy.

  9. Absolute neutrophil count ≥1500/µL, platelet ≥100000/mm3, hemoglobin ≥10g/dL

Exclusion Criteria:

* 1. Prior treatment with any CDK4/6 inhibitor.

  2. Inflammatory or stage IV or bilateral breast cancer.

  3. History of allergic reactions caused by chemical or biological components similar to CDK4/6 inhibitors.

Patients who received any drugs or substances that were effective CYP3A isoenzyme inhibitors or inducers within 7 days of enrollment.

5. Uncontrolled coexisting medical conditions may limit adherence to study requirements.

6. Pregnant women with a negative pregnancy test within 14 days before admission or women of childbearing potential.

7. Patients with a history of any malignancy were not eligible.

8. Patients receiving endocrine therapy within 5 years before diagnosis of current malignancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 weeks
  ORR is defined as proportion of patients demonstrating either a partial response (PR) or a complete response (CR)

SECONDARY OUTCOMES:
change in Ki67 | up to 24 weeks
  change in Ki67 from baseline to end of treatment
complete cell cycle arrest | up to 4 weeks
  The proportion of patients with Ki-67≤2.7% on day 15 of cycle 1 treatment
Invasive disease free survival（iDFS） | up to 3 years
  Time from adjuvant therapy to disease recurrence in patients with invasive disease

CONTACTS AND LOCATIONS:
Locations (1):
- No. 119 Zhuodaoquan South Road, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No